CLINICAL TRIAL: NCT00290589
Title: Utility of Intramuscular Corticosteroids for Radicular Low Back Pain
Brief Title: A Trial of Corticosteroids for Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, Prof. Emergency Medicine, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03-05-107
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Radicular Low Back Pain
Keywords: low back pain; emergency department; corticosteroids
MeSH Terms: conditions — Low Back Pain; Emergencies | interventions — Steroids; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes

ARMS (2):
- Intramuscular methylprednisolone acetate (Experimental): Methylprednisolone acetate 160mg intramuscular injection
  Interventions: Drug: Intramuscular methylprednisolone acetate
- Placebo (Placebo Comparator): Placebo intramuscular injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intramuscular methylprednisolone acetate — Intramuscular methylprednisolone acetate 160mg
  Other Names: steroid
  Arms: Intramuscular methylprednisolone acetate
Drug: Placebo — Normal saline intramuscular injection
  Other Names: saline solution
  Arms: Placebo

SUMMARY:
Low back pain is a common symptom that functionally disables many people. When the low back pain is accompanied by pain that shoots down the leg, it is felt to be caused by a herniated disc. We are conducting this study to determine if a powerful anti-inflammatory agent will decrease the pain and functional impairment that is associated with this illness.

DETAILED DESCRIPTION:
This is a randomized, double-blind placebo-controlled clinical trial evaluating intramuscular methylprednisolone acetate as adjunctive therapy for radicular low back pain. This trial randomizes subjects after they had been evaluated and treated in the ED and are ready for discharge. All subjects are followed by telephone call one week and one month after ED discharge. In addition to the steroid injection, all subjects are given a complimentary one week supply of naproxen 500 mg tablets and oxycodone 5mg/ acetaminophen 325 tablets and a detailed low back pain instruction sheet. This study was approved by the Montefiore Medical Center institutional review board.

Patients are included if their low back pain lasted less than one week, if they are 50 years old or younger, and if they had not experienced any direct trauma to the back during the previous week. Low back pain is described as pain originating below the tips of the scapulae and above the buttocks.Patients are only included if their straight leg raise test, as described below, is positive. Patients are excluded if the emergency physician felt that there is a high likelihood that the patient has a secondary cause of low back pain, e.g., metastatic bone disease or infection. Patients are also excluded for temperature greater than 100.3 degrees, pregnancy, lactation, allergy to or intolerance of a study medication. Patients can only enroll once. Patients can not have had another episode of back pain within four weeks prior to the current back pain attack. Patients are excluded for systemic steroid use within four weeks, a history of back surgery, a neoplasia known to metastasize, a chronic pain syndrome, an inflammatory arthritis, suspected vascular, urologic or gynecologic pathology, or direct blunt trauma to the back within the previous week.

Rationale for the straight leg raise test: Although the true test characteristics of the straight leg raise test are unknown, a positive ipsilateral straight leg raise is felt to be a sensitive marker for a herniated intervertebral disc. Therefore, if this test is negative, it can help rule-out the disease. To maintain a homogenous cohort, subjects were stratified based on results of the straight leg raise test. Many definitions of the straight leg raise test exist. In order to identify distinct populations, the research assistants were given a strictly-defined, conservative definition of this test: namely, the test was considered positive if a subject had ipsilateral pain shooting below the knee when either leg was raised between 30 and 70 degrees, as measured with a protractor. Contralateral pain below the knee, considered more specific for a herniated disc, was also considered a positive straight leg raising test.

All patients with low back pain are treated at the discretion of the attending physician. When the patient's pain had been controlled to a level sufficient for the patient to be discharged, the patient is asked for consent to participate as a research subject. After consent is obtained, subjects receive an intramuscular injection of methylprednisolone acetate or placebo. All subjects are discharged with a "back pack" containing 14 tablets of naproxen 500mg, 12 tablets of oxycodone 5mg/ acetaminophen 325 tablets, and a standardized discharge instruction sheet.

Subjects are followed-up by telephone at one week and one month after discharge. At each of these telephone interviews, research assistants read standardized questions about pain and activity limitations from the data collection instrument.

ELIGIBILITY:
Inclusion Criteria:

* 21-50 years old, non-traumatic low back pain for one week or less,

Exclusion Criteria:

* fever, pregnancy, lactation, allergy or intolerance to study medication, suspected active oncologic, urologic, or gynecologic disease

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2003-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Friedman, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intramuscular Methylprednisolone Acetate | Placebo
Started | 39 | 43
Completed | 37 | 41
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intramuscular Methylprednisolone Acetate | Placebo | Total
Number analyzed (Participants) | 39 | 43 | 82
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39 (9) | 37 (8) | 38 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 18 | 21 | 39
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 43 | 82
Duration of Back Pain Prior to Study [Mean (Inter-Quartile Range); unit: hours] | 48 [24 to 72] | 48 [14 to 72] | 48 [24 to 72]

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale (0-10), an Interval Pain Scale, on Which 0 Indicates no Pain and 10 Indicates the Worst Pain Imaginable
Description: Improvement in Numerical Rating Scale between the time of the emergency department visit and the one month telephone call is rated on an 11-point scale ranging from 0-10 with 0 indicating no pain and 10 indicating worse pain imaginable.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intramuscular Methylprednisolone Acetate | Placebo
Number analyzed (Participants) | 39 | 43
units on a scale | 7.1 (3.0) | 5.8 (3.5)

2. Primary Outcome: Functional Disability Scales
Description: The low back pain functional disability scale is the Roland Morris Disability questionnaire score (RMDQ). The RMDQ is a 24-item low back pain functional scale recommended for use in low back pain research.Higher scores signify greater low back-related functional impairment.0= no functional impairment, 24= severe functional impairment.
Time Frame: 1 month
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Intramuscular Methylprednisolone Acetate | Placebo
Number analyzed (Participants) | 39 | 43
units on a scale | 0 [0 to 0] | 0 [0 to 11]

3. Secondary Outcome: Number of Patients Using Analgesics
Description: Use of analgesics for low back pain (within the previous 24 hours)
Time Frame: Assessed at 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intramuscular Methylprednisolone Acetate | Placebo
Number analyzed (Participants) | 37 | 40
Participants | 8 | 17

ADVERSE EVENTS:
Arm/Group | Intramuscular Methylprednisolone Acetate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/41
Other Adverse Events (participants affected / at risk) | 12/37 | 10/43
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intramuscular Methylprednisolone Acetate (N=37) | Placebo (N=43)
Drowsiness (General disorders) | 6 (6) | 5 (43)
Stomach Pain (Gastrointestinal disorders) | 4 (4) | 2 (43)
Mood Change (Nervous system disorders) | 1 (1) | 0 (0)
Bloating (Gastrointestinal) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Other (General disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes